CLINICAL TRIAL: NCT01652391
Title: Modulation of Cognitive Control in Healthy and Depressed Subjects by Transcranial Direct Current Stimulation
Brief Title: Modulation of Cognitive Control by Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Professer, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 211/2010BO1_1
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal transcranial direct current stimulation (Experimental): Anodal transcranial direct current stimulation (tDCS) 20min, 1mA, F3 (EEG 10/20), reference right M. deltoideus
  Interventions: Device: Transcranial direct current stimulation (tDCS); DC-STIMULATOR (NeuroConn GmbH, Ilmenau, Germany)
- Sham transcranial direct current stimulation (Sham Comparator): Sham transcranial direct current stimulation (tDCS) 40s, 1mA, F3 (EEG 10/20), reference right M. deltoideus
  Interventions: Device: Transcranial direct current stimulation (tDCS); DC-STIMULATOR (NeuroConn GmbH, Ilmenau, Germany)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS); DC-STIMULATOR (NeuroConn GmbH, Ilmenau, Germany)

SUMMARY:
Insufficient cognitive control over emotional distracters is characteristic for major depressive disorder (MDD). Hypoactivation of the dorsolateral prefrontal cortex (dlPFC) is associated with this deficit. In this study the investigators assess the effect of an enhancement of dlPFC activity in MDD patients by anodal transcranial direct current stimulation (tDCS) on cognitive control.

In a double-blinded, balanced randomized, sham-controlled crossover trial the investigators determine the effect of a single-session tDCS to the left dlPFC on cognitive control in MDD patients and healthy controls. To assess the cognitive control the investigators use a delayed response working memory (DWM) task with pictures of varying valence presented during the delay period.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* informed consent
* in the patients group: Major depressive disorder, no antidepressant medication or stability over 1 week

Exclusion Criteria:

* seizures
* cardiac pacemaker
* deep brain stimulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Correctness of response | The primary outcome measure is obtained during the intervention (20min tDCS or sham stimulation).

SECONDARY OUTCOMES:
Reaction time | The secondary outcome measure is obtained during the intervention (20min tDCS or sham stimulation).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitiy Hospital Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Wolkenstein L, Plewnia C. Amelioration of cognitive control in depression by transcranial direct current stimulation. Biol Psychiatry. 2013 Apr 1;73(7):646-51. doi: 10.1016/j.biopsych.2012.10.010. Epub 2012 Dec 6. PMID 23219367